CLINICAL TRIAL: NCT00939237
Title: Trial of Ateronon for Carotid Atherosclerosis and Biomarkers in Patients With Stable Coronary Heart Disease
Brief Title: Trial of Lycopene/Ateronon for Secondary Prevention of Coronary Heart Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: CamNutra Ltd. (Industry); Cambridge Theranostics Ltd (Industry)
Responsible Party: Principal Investigator, Howard D. Sesso, ScD, MPH, Associate Epidemiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-P-000202 BWH
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Heart Disease
Keywords: Coronary heart disease; Carotid intima-media thickness; Biomarkers
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Ateronon (Experimental): 7 mg lycopene dietary supplement supplied as one Ateronon capsule taken daily
  Interventions: Drug: Ateronon
- Placebo (Placebo Comparator): placebo dietary supplement supplied as one capsule taken daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ateronon — 7 mg lycopene dietary supplement supplied as one Ateronon capsule taken daily
  Arms: Active Ateronon
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Ateronon, a nutritional supplement that contains lycopene from tomatoes has a favorable effect on carotid atherosclerosis, lipid levels, and other biomarkers of coronary heart disease.

The trial was stopped early due to insufficient financial support from the initial study collaborator, Cambridge Theranostics Ltd. Collected patient data are sufficient for final trial-based analyses to be conducted with financial support from the new study collaborator, CamNutra Ltd. The data will still be analyzed according to the original study aims.

DETAILED DESCRIPTION:
Lycopene, a carotenoid mainly found in tomato-based food products, has strong antioxidant properties relative to other carotenoids and has been postulated to play a role in the prevention of coronary heart disease through a variety of mechanisms. Lycopene cooked and consumed in oil mediums is optimal for not only its efficient absorption, but also its potential clinical effectiveness. Studies have also linked serum lycopene with the early stages of atherosclerosis, as measured by carotid artery intima-media thickness (IMT), a noninvasive ultrasound examination of the carotid arteries and potential surrogate endpoint for subsequent cardiovascular morbidity and mortality used in previous clinical trials of vitamin supplements. Short-term intervention studies of lycopene supplements are limited, having explored mechanisms through which lycopene or its readily absorbable food sources may increase plasma lycopene or induce changes in other relevant biochemical markers impacting the subsequent risk of coronary heart disease. Ateronon is a lycopene supplement developed with the understanding that the potential clinical effectiveness of lycopene is impacted by its bioavailability. A single daily 7 mg tablet of Ateronon provides more bioavailable lycopene than diet alone, is absorbed efficiently, and completely inhibits the atherogenic lipid oxidation processes in subjects. Clinical studies suggest that short-term treatment with Ateronon among those with coronary heart disease leads to favorable reductions in lipid levels, lipoprotein oxidation, blood pressure, and Rose-Blackburn scores. Therefore, we will conduct a randomized, double-blind, placebo-controlled clinical trial of 7 mg Ateronon taken daily for 1 year among 200 patients aged ≥50 years with stable coronary heart disease. This clinical trial is a collaborative effort between the Division of Preventive Medicine and the Vascular Medicine Program in the Division of Cardiology. Our primary aim is whether taking Ateronon for 1 year is associated with favorable changes in carotid IMT. Secondary aims expand to whether Ateronon leads to favorable 1-year changes in coronary biomarkers related to oxidative stress and endothelial dysfunction; blood pressure; plasma carotenoids; AtheroAbzyme levels; and other traditional coronary biomarkers. This clinical trial of Ateronon seeks to improve our understanding of various mechanisms through which Ateronon, a concentrated and highly bioavailable form of lycopene, may reduce the risk of developing coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Brigham and Women's Hospital Cardiology Clinic patients with history of coronary heart disease occurring at least 6 months ago:

  * history of myocardial infarction (MI) confirmed by medical records AND/OR
  * history of percutaneous coronary intervention (PCI) or coronary artery bypass surgery (CABG)
* Compliance during run-in as demonstrated by taking at least 66% of study medications
* Ability and willingness to complete questionnaires concerning medical history, concomitant medication use, coronary heart disease risk factors, potential adverse events, and diet

Exclusion Criteria:

* History of carotid stent, carotid endarterectomy, or carotid artery surgery
* History of diagnosed congestive heart failure meeting New York Association Functional Classification III or IV criteria
* Any initiation or change in statin use or other lipid-lowering treatment within 3 months of randomization
* Lactose intolerance
* Allergies to whey protein
* Allergies to soy protein
* History of active cancer diagnosis (except non-melanoma skin cancer) within last 3 years
* Life expectancy < 1 year
* Women who are pregnant, nursing, or intend pregnancy during the period of treatment
* Plan to relocate out of Boston area within the next year
* Inability to provide informed consent
* Carotid artery occlusion or dissection at baseline carotid IMT assessment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Carotid intima-media thickness | Baseline, 6 months, and 12 months

SECONDARY OUTCOMES:
Biomarkers for coronary heart disease | Baseline, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Howard D. Sesso, ScD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States